CLINICAL TRIAL: NCT06064331
Title: Effect of Intravenous Lignocaine Infusion on Intraoperative End Tidal Desflurane Concentration Requirements: A Randomised Double-Blinded Controlled Study
Brief Title: Effect of Intravenous Lignocaine Infusion on Intraoperative End Tidal Desflurane Concentration Requirements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FF-2021-024
Record Dates: First submitted 2022-06-15; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Cholelithiases; Appendicitis; Ovarian Cysts
Keywords: Lignocaine; Desflurane
MeSH Terms: conditions — Cholelithiasis; Appendicitis; Ovarian Cysts | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Lignocaine (Experimental): Group Lignocaine will receive an IV bolus dose of 1.5 mg/kg of 2% lignocaine HCL diluted up to 10 ml with normal saline in a 10 ml syringe which will be delivered via a syringe pump over a period of 3 min. This is then followed by an IV infusion at the rate of 1 mg/kg/h of 2% lignocaine HCL in a 20 ml syringe which will be administered by another syringe pump.
  Interventions: Drug: Lignocaine
- Group Placebo (Placebo Comparator): Patients in Placebo Group will receive an IV bolus of 10 ml of normal saline over a period of 3 min followed by an IV infusion of an equal volume of normal saline, both of which will be delivered by separate syringe pumps.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lignocaine — IV bolus of 1.5 mg/kg of lignocaine 2% diluted in 10 ml syringe over 3 mins followed by infusion at 1 mg/kg/h of lignocaine 2% in 20 ml syringe
  Arms: Group Lignocaine
Drug: Placebo — IV bolus of 10 ml normal saline over 3 min followed by infusion of equal volume of normal saline in 20 ml syringe
  Arms: Group Placebo

SUMMARY:
Lignocaine is a local anaesthetic that is widely used in all medical and surgical fields. Many clinical studies have shown that intravenous (IV) lignocaine given in the perioperative period was safe, reduced airway complications, obtunds cough reflex, reduce sore throat, pain, opioid consumption, nausea, length of hospital stay. Multiple animal studies have shown that IV lignocaine was able to lower anaesthetic gas requirements. Desflurane is an anaesthetic gas that has a rapid onset and offset of action. This study aims to evaluate the effect of IV lignocaine infusion on desflurane requirements.

Hypothesis of the study is that IV lignocaine infusion reduces desflurane requirements.

DETAILED DESCRIPTION:
All volunteers will be randomly assigned into two groups based on computer generated randomisation tables.

Group Lignocaine will receive an IV bolus dose of 1.5 mg/kg of 2% lignocaine HCL diluted up to 10 ml with normal saline in a 10 ml syringe which will be delivered via a syringe pump over a period of 3 min. This is then followed by an IV infusion at the rate of 1 mg/kg/h of 2% lignocaine HCL in a 20 ml syringe which will be administered by another syringe pump.

Group Placebo will receive an IV bolus of 10 ml of normal saline over a period of 3 min followed by an IV infusion of an equal volume of normal saline, both of which will be delivered by separate syringe pumps.

After induction of anaesthesia, all volunteers will be ventilated with Aisys™ CS² anaesthesia machine. Anaesthesia shall be maintained with desflurane, in 50% oxygen-air balance with a total flow of 1.0 L/min. The end tidal desflurane (Et-Des) concentration will be adjusted to maintain a target BIS of between 40-60.

Desflurane and study infusions will be discontinued and estimation of desflurane cost and volume used will be estimated at the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anaesthesiology (ASA) I or II patients.
2. Patients aged between 18-75 years of age.
3. Patients scheduled for elective laparoscopic cholecystectomy.
4. Patients scheduled for laparoscopic hernioplasty.
5. Patients scheduled for emergency laparoscopic appendicectomy.
6. Patients scheduled for emergency laparoscopic cystectomy.
7. Patient weight ranging from 50 - 100 kg.
8. Surgery lasting at least one hour.

Exclusion Criteria:

1. Patients with a known allergy to study drug.
2. Patients with body mass index (BMI) more than 35 kg m-2.
3. Patients who are taking sedatives.
4. Patients with chronic substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
End Tidal Desflurane at Bispectral Index (BIS) 40-60 | Intraoperatively until surgery ends
  Percentage of reduction in end tidal desflurane between Lignocaine Group Versus Placebo Group
Volume of Desflurane used to maintain BIS 40-60 | Intraoperatively until surgery ends
  Percentage of reduction of desflurane volume required during surgery between Lignocaine Group Versus Placebo Group
Cost of Desflurane used to maintain BIS 40-60 | Intraoperatively until surgery ends
  Percentage of reduction of cost of desflurane between the 2 groups

SECONDARY OUTCOMES:
Systolic, diastolic and mean arterial pressure (mmHg) intraoperatively | Intraoperatively until surgery ends
  Systolic, diastolic and mean arterial pressure(mmHg) intraoperatively will be recorded and compared between the two groups
Heart rate (beats per minute) intraoperatively | Intraoperatively until surgery ends
  Heart rate (bpm) intraoperatively will be recorded and compared between the two groups
Opioid usage (mcg/kg) | Intraoperatively until surgery ends
  Incidence of patients require rescue opioid (mcg/kg) intraoperatively and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Syarifah Noor Nazihah Sayed Masri, MD, Principal Investigator — National University of Malaysia
Locations (1):
- Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 5 years within study period
Access Criteria: Registered with clinicaltrials.gov

REFERENCES:
- [Background] Weinberg L, Jang J, Rachbuch C, Tan C, Hu R, McNicol L. The effects of intravenous lignocaine on depth of anaesthesia and intraoperative haemodynamics during open radical prostatectomy. BMC Res Notes. 2017 Jul 6;10(1):248. doi: 10.1186/s13104-017-2570-4. PMID 28683817
- [Background] Yang SS, Wang NN, Postonogova T, Yang GJ, McGillion M, Beique F, Schricker T. Intravenous lidocaine to prevent postoperative airway complications in adults: a systematic review and meta-analysis. Br J Anaesth. 2020 Mar;124(3):314-323. doi: 10.1016/j.bja.2019.11.033. Epub 2020 Jan 28. PMID 32000978
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Kuo CP, Jao SW, Chen KM, Wong CS, Yeh CC, Sheen MJ, Wu CT. Comparison of the effects of thoracic epidural analgesia and i.v. infusion with lidocaine on cytokine response, postoperative pain and bowel function in patients undergoing colonic surgery. Br J Anaesth. 2006 Nov;97(5):640-6. doi: 10.1093/bja/ael217. Epub 2006 Sep 4. PMID 16952918
- [Background] Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, Hering W. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesth Analg. 2004 Apr;98(4):1050-1055. doi: 10.1213/01.ANE.0000104582.71710.EE. PMID 15041597
- [Background] Reed R, Doherty T. Minimum alveolar concentration: Key concepts and a review of its pharmacological reduction in dogs. Part 2. Res Vet Sci. 2018 Jun;118:27-33. doi: 10.1016/j.rvsc.2018.01.009. Epub 2018 Feb 2. PMID 29421482
- [Background] Acevedo-Arcique CM, Ibancovichi JA, Chavez JR, Gutierrez-Blanco E, Moran-Munoz R, Victoria-Mora JM, Tendillo-Cortijo F, Santos-Gonzalez M, Sanchez-Aparicio P. Lidocaine, dexmedetomidine and their combination reduce isoflurane minimum alveolar concentration in dogs. PLoS One. 2014 Sep 18;9(9):e106620. doi: 10.1371/journal.pone.0106620. eCollection 2014. PMID 25232737
- [Background] Rezende ML, Wagner AE, Mama KR, Ferreira TH, Steffey EP. Effects of intravenous administration of lidocaine on the minimum alveolar concentration of sevoflurane in horses. Am J Vet Res. 2011 Apr;72(4):446-51. doi: 10.2460/ajvr.72.4.446. PMID 21453144
- [Background] Pypendop BH, Ilkiw JE. The effects of intravenous lidocaine administration on the minimum alveolar concentration of isoflurane in cats. Anesth Analg. 2005 Jan;100(1):97-101. doi: 10.1213/01.ANE.0000139350.88158.38. PMID 15616060
- [Background] Kapoor MC, Vakamudi M. Desflurane - revisited. J Anaesthesiol Clin Pharmacol. 2012 Jan;28(1):92-100. doi: 10.4103/0970-9185.92455. PMID 22345954
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT06064331/Prot_SAP_ICF_000.pdf